CLINICAL TRIAL: NCT00005702
Title: Promoting Smoking Cessation in Hospital Patients
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4302; R01HL054132 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To experimentally test methods to promote long-term smoking cessation in hospitalized patients.

DETAILED DESCRIPTION:
BACKGROUND:

Cigarette smoking is a vitally important public health problem. It is a major contributor to cardiovascular disease and one of the leading causes of cancer and respiratory disease. Research in primary care over the last two decades has indicated that smoking cessation interventions in medical settings can be effective. However, there have been few published reports of research examining the effectiveness of smoking cessation interventions in hospital settings. In-patient smoking cessation interventions can potentially reach a large number of smokers. A hospital stay can also be an effective "teachable moment" for smoking cessation advice. Smoking bans in place in hospitals make it a time of enforced abstinence and therefore, an opportunity to overcome the symptoms of physical addiction. Patients are removed from their usual environmental cues for smoking, making initial cessation easier, and they might be particularly receptive to preventive health messages at a time of ill-health. Finally, there is increased access to health care providers whom patients see as valid and knowledgeable sources of health information.

DESIGN NARRATIVE:

All smokers admitted to three hospitals over a 27-month period were identified as part of the admissions process. Those who met eligibility requirements were randomly assigned to one of three treatment conditions: minimal care; a low intensity intervention whose centerpiece was brief firm advice by health care providers and labelling of the smokers' charts (PA intervention); and the PA intervention plus more intensive counseling and follow-up after discharge performed by a research nurse (PA+NC intervention). Intervention components included provision of smoking cessation manuals and training of health care providers (all conditions); structural reminders to health care providers to give smoking cessation advice and provision of smoking cessation advice by a variety of health care providers on several different occasions (PA and PA+NC); and in-hospital counseling tailored to patient characteristics, feedback about a biological marker of smoking, a stepped care approach, and follow-up telephone counseling after discharge (PA+NC only). All participants were followed for twelve months after discharge from the hospital to examine the relative effectiveness and cost-effectiveness of the smoking cessation programs. In addition, information about smoking cessation advice given to study patients by primary care physicians in the twelve months after discharge from hospital was gathered to assess the possible synergistic effects of advice provided in in-patient and out-patient settings.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-05; Study Completion 2000-04

REFERENCES:
- [Background] Nicholson JM, Hennrikus DJ, Lando HA, McCarty MC, Vessey J. Patient recall versus physician documentation in report of smoking cessation counselling performed in the inpatient setting. Tob Control. 2000 Dec;9(4):382-8. doi: 10.1136/tc.9.4.382. PMID 11106707
- [Background] McCarty MC, Zander KM, Hennrikus DJ, Lando HA. Barriers among nurses to providing smoking cessation advice to hospitalized smokers. Am J Health Promot. 2001 Nov-Dec;16(2):85-7, ii. doi: 10.4278/0890-1171-16.2.85. PMID 11727593
- [Background] McCarty MC, Hennrikus DJ, Lando HA, Vessey JT. Nurses' attitudes concerning the delivery of brief cessation advice to hospitalized smokers. Prev Med. 2001 Dec;33(6):674-81. doi: 10.1006/pmed.2001.0944. PMID 11716666